CLINICAL TRIAL: NCT01332474
Title: BOTOX®(BOTOX is a Registered Trade Mark of Allergan, Inc) Injection 50 and 100 Treatment of Equinus Foot Due to Lower Limb Spasticity in Juvenile Cerebral Palsy Patients Aged 2-year or Older: Investigation of Patient Background Characteristics
Brief Title: JCP Study of Investigation of Patient Background Characteristics
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114324
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Spasticity, Post-Stroke
Keywords: Botox; JCP
MeSH Terms: conditions — Muscle Spasticity | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- JCP: treatment of Equinus Foot due to Lower Limb Spasticity in Juvenile Cerebral Palsy Patients Aged 2-year or Older
  Interventions: Drug: BOTOX

INTERVENTIONS:
Drug: BOTOX — BOTOX

SUMMARY:
To collect the background characteristics of juvenile cerebral palsy patients aged 2-year or older prescribed BOTOX for the treatment of equines foot due to lower limb spasticity, compare them with those of patients whose deaths or adverse drug reactions (ADRs) related to the possible spread of toxin are reported through the spontaneous ADR reporting system, and discuss potential risk factors for such ADRs.

DETAILED DESCRIPTION:
1. In each of prospective medical institutions (where BOTOX is expected to be prescribed annually to at least 10 juvenile cerebral palsy patients aged 2-year or older), the Medical Representative will explain the objectives, subjects and methods of the investigation to the prospective investigator (i.e., a physician who will prescribe BOTOX and can comply with the protocol of the investigation) and ask for his/her participation in the investigation.
2. When the physician agrees to participate in the investigation, a written agreement will be concluded between GSK and the head (e.g. director) of the medical institution prior to the start of the investigation.
3. After the completion of the investigation period, the physician will complete the case report form (CRF) for the patients prescribed BOTOX by him/her during the investigation period. The information of the patients who developed ADRs will be collected separately through the spontaneous ADR reporting system on a daily basis.

ELIGIBILITY:
Inclusion Criteria:

* Background factors:

The following background characteristics will be compared between the patients collected during the investigation and the patients whose deaths or ADRs related to the possible spread of toxin are reported through the spontaneous ADR reporting system, to discuss the potential risk factors for death or spread of toxin:

1. severity of indication (cerebral palsy) prior to use of BOTOX
2. Medical history/concurrent medical conditions (e.g., dysphagia, seizure, pulmonary disorder, neuromuscular disorder, and cardiac disorder, and others) ; Yes/No, and if yes, specify the diseases
3. Use of concomitant drugs and non-drug therapies
4. Dose per kg body weight
5. Dose per injection site (e.g., gastrocnemius muscle, soleus muscle, tibialis posterior muscle)

Exclusion Criteria:

* patients whose adverse drug reactions (ADRs)

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients aged 2-year or older
Sampling Method: Probability Sample
Enrollment: 326 (Actual)
Dates: Start 2010-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
compare JCP patients with those of patients whose deaths or adverse drug reactions (ADRs) related to the possible spread of toxin are reported through the spontaneous ADR reporting system. | 2010/5/1-2010/8/31

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline